CLINICAL TRIAL: NCT05763069
Title: The HOME Study: Home Monitoring of High-risk Pregnancies
Brief Title: HOME: Home Monitoring of High-risk Pregnancies
Status: Enrolling by invitation | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian SIDS and Stillbirth Society (Other); University of Oxford (Other); Rigshospitalet, Denmark (Other); Sykehuspartner (Unknown); Dignio (Unknown); Medexa (Unknown)
Responsible Party: Principal Investigator, Anne Cathrine Staff, Professor, Head of research, MD; PhD, Oslo University Hospital
Other Study IDs: 473099
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hypertensive Disorder of Pregnancy; Premature Preterm Rupture of Membranes; Preeclampsia; High Risk Pregnancy; Previous Adverse Obstetric Outcome
MeSH Terms: conditions — Toxemia; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home surveillance of pregnancies at risk — Offer women with pregnancies at risk home surveillance instaed of more frequent hospital out-patient visits and/or hospitalisation: cardiotocographia (CTG), patient measurements of CRP, temperature, blood pressure, and clinical signs of infection or severe forms of preeclampsia.

SUMMARY:
High-risk pregnancies often require long-term hospitalization or outpatient maternal and/or fetal monitoring, placing a burden on patients, hospital resources and society. The demand for intensified pregnancy surveillance and interventions is increasing, due to the increased prevalence of risk factors like obesity and advanced maternal age, as well as altered guidelines resulting in increasing labor induction rates.The main aims of the HOME study (Home monitoring of pregnancies at risk) are to assess if home monitoring of selected high-risk pregnancies for maternal and fetal wellbeing is feasible, safe (in a clinical trial), cost-efficient, and simultaneously empowers the users.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia
* Gestational Hypertension
* Premature Preterm Rupture of Membranes
* High Risk Pregnancy
* Previous adverse obstetric outcomes

Exclusion Criteria:

* Multiples (twins, triplets etc)
* Patient or fetus in immediate need for delivery
* Not understanding Norwegian
* Not mastering the technological aspects of home monitoring
* Long travel distance to Obstetric Department

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women identified with the at-risk pregnancies described above, attending Oslo University Hospital's Department of Obstetrics (some controls will also be recruited at another South-Eastern Norway Dept of Obstetrics, at Drammen hospital).
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Home monitoring of high-risk pregnancies | 2022-2035
  Development of secure data transfer systems from home to electronic patient records at the hospital

SECONDARY OUTCOMES:
User acceptability of home monitoring | 2022-2035
  Patient expectations (prior to intervention) and reported acceptability and quality of life
Clinical safety of home monitoring | 2022-2035
  Non-inferior compared to patients not undergoing home monitoring ("controls")
Health economics of home monitoring | 2022-2035
  Non-inferior compared to health economics in patients not undergoing home monitoring ("controls")
Placenta-associated biomarkers: improving CTG prediction of adverse outcomes? | 2023-2035
  Do placenta-associateed circulating biomarkers prior to delivery, used in an algoritm, improve CTG-assisted prediction of fetal asphyxia?

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cathrine Staff, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Pending on patient consent and ethical approval details

REFERENCES:
- [Derived] Waldum AH, Pay ASD, Aasbo G, Mishra VK, Sugulle M, Staff AC. The HOME (home monitoring of high-risk pregnancies) study: a study protocol for an observational study of a telemedicine-assisted follow-up at home vs. hospitalization. Front Glob Womens Health. 2025 Jul 14;6:1599153. doi: 10.3389/fgwh.2025.1599153. eCollection 2025. PMID 40726590